CLINICAL TRIAL: NCT04235101
Title: A Two-part Phase I Study With the Antibody-drug Conjugate SYD985 in Combination With Niraparib to Evaluate Safety, Pharmacokinetics and Efficacy in Patients With HER2-expressing Locally Advanced or Metastatic Solid Tumors.
Brief Title: Phase I Study of SYD985 With Niraparib in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Byondis B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYD985.004
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor
Keywords: Solid Tumor; Anti-body Drug Conjugate; ADC; niraparib
MeSH Terms: interventions — trastuzumab duocarmazine; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYD985 + Niraparib (Experimental): SYD985, Intravenous, every 3 weeks (Q3W) Niraparib taken orally and either 100 mg, 200 mg or 300 mg once daily for either 1, 2 or 3 weeks.
  Interventions: Drug: SYD985 + Niraparib

INTERVENTIONS:
Drug: SYD985 + Niraparib — SYD985 powder for concentrate for solution for infusion Niraparib 100 mg per hard capsule
  Other Names: (vic-)trastuzumab duocarmazine + Zejula

SUMMARY:
SYD985.004 is a two-part phase I study with the antibody-drug conjugate SYD985 in combination with niraparib aimed at evaluating safety, pharmacokinetics and efficacy in patients with HER2-expressing locally advanced or metastatic solid tumours.

DETAILED DESCRIPTION:
This is an open-label, single-arm study in which patients with HER2-expressing locally advanced or metastatic solid tumours will be treated with both an anti-body drug conjugate SYD985 and a Poly (ADP-ribose) Polymerase (PARP) inhibitor niraparib. SYD985 is an antibody-drug conjugate and consists of two parts. The antibody part binds to a protein that exists on different types of cancer cells (HER2 protein). When SYD985 binds to this protein, it will be taken up by the cancer cell. The second part of the drug, a toxin, will be cleaved in the cell and subsequently kills the cancer cell. Niraparib blocks the action of enzymes PARP-1 and PARP-2, which help to repair damaged DNA in cells when the cells divide to make new cells. By blocking PARP enzymes, the damaged DNA in cancer cells cannot be repaired, and, as a result, the cancer cells die.

Part 1 includes patients with locally advanced or metastatic HER2-expressing solid tumours of any origin that showed progression on standard therapy or for whom no standard therapy exists. Patients will receive SYD985 infusions every three weeks in combination with niraparib until progression of the cancer or unacceptable toxicity develops. In this first part of the study, different doses of niraparib will be given for either 1, 2 or 3 weeks.

Part 2 includes patients with advanced or metastatic breast, ovarian or endometrial cancer that showed progression on standard therapy or for whom no standard therapy exists. Patients will receive SYD985 infusions every three weeks in combination with niraparib until progression of the cancer or unacceptable toxicity develops.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age ≥ 18 years at the time of signing first informed consent;
* Patient with a histologically-confirmed, locally advanced or metastatic tumour who has progressed on standard therapy or for whom no standard therapy exists, with the following restriction:

  * Part 1: solid tumours of any origin;
  * Part 2: breast cancer, ovarian cancer or endometrial carcinoma/carcinosarcoma;
* HER2 tumor status at least 1+ as assessed by immunohistochemistry (IHC) as determined by the local laboratory;
* Presence of a tumor lesion accessible for biopsy and patient should be willing to undergo a fresh biopsy for central HER2 testing and genetic testing, unless adequate (biopsy) tumour material is available obtained < 6 months prior to signing the main informed consent;
* At least one measurable cancer lesion as defined by the Response Evaluation Criteria for Solid Tumours (RECIST version 1.1);
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1;
* Adequate organ function.

Exclusion Criteria:

* Having been treated with:

  1. DUBA-containing ADCs at any time;
  2. Anthracycline treatment within 8 weeks prior to start of study treatment;
  3. Other anticancer therapy including chemotherapy, immunotherapy, or investigational agents within 4 weeks prior to start of study treatment or 5 times the half-life of the therapy, whichever is shorter;
  4. Radiotherapy within 4 weeks prior to start of study treatment or within 1 week for palliative care (as long as the lungs were not exposed);
  5. Hormone therapy within 1 week prior to start of study treatment. The patient must have sufficiently recovered from any treatment-related toxicities to NCI CTCAE Grade ≤ 1 (except for toxicities not considered a safety risk for the patient at the investigator's discretion);
* History or presence of keratitis;
* Left ventricular ejection fraction (LVEF) < 50% as assessed by either echocardiography or multigated acquisition (MUGA) scan at screening, or a history of clinically significant decrease in LVEF during previous trastuzumab containing treatment leading to permanent discontinuation of treatment;
* History (within 6 months prior to start of study treatment) or presence of clinically significant cardiovascular disease such as unstable angina, congestive heart failure, myocardial infarction, uncontrolled hypertension, or cardiac arrhythmia requiring medication;
* History or presence of idiopathic pulmonary fibrosis, organizing pneumonia (e.g. bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan;
* Severe, uncontrolled systemic disease (e.g. clinically significant cardiovascular, pulmonary, or metabolic disease) at screening;
* Symptomatic brain metastases, brain metastasis requiring steroids to manage symptoms or treatment for brain metastases within 8 weeks prior to start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | 21 days
  First cycle

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 2 years
Area under the plasma concentration versus time curve (AUC) of SYD985 and niraparib | Baseline, Days 1,8,15 of Cycle 1, Days 1,8,15 of Cycle 2, Day 1 of subsequent cycles up to 6 months
Peak plasma concentration of SYD985 and niraparib | Baseline, Days 1,8,15 of Cycle 1, Days 1,8,15 of Cycle 2, Day 1 of subsequent cycles up to 6 months
Change from baseline in hematology and blood chemistry parameters | Baseline and every cycle up to 2 years
Number of patients with antibodies against SYD985 | Baseline and every cycle up to 2 years
Objective response rate | Baseline and every two cycles for up to 6 months, subsequent every 4 cycles up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Koper, Study Director — Byondis B.V., The Netherlands
Locations (6):
- Belgium (2):
  - University Hospital Antwerp, BE, Antwerp
  - Institut Jules Bordet, Brussels
- Radboud University Medical Center/ NL, Nijmegen, Netherlands
- United Kingdom (3):
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust/ UK, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust/UK, Newcastle

IPD SHARING:
Plan to Share IPD: No